CLINICAL TRIAL: NCT02892032
Title: Mobile Based Attention Bias Modification Training for Chronic Pain
Brief Title: Attention Training Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Joel Katz, Professor. Canada Research Chair in Health Psychology., York University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: e2016-240
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Modification Training (Experimental): ABMT is a newly emerging intervention that trains patients to override their tendency to focus on threatening aspects of an event and to interpret events as more neutral and therefore less stressful
  Interventions: Behavioral: Attention Modification Training
- No Attention Modification Training (Placebo Comparator): There is no disengagement of attention from a target stimulus. Attention is divided equally between two stimuli on the screen.
  Interventions: Behavioral: No Attention Modification Training

INTERVENTIONS:
Behavioral: Attention Modification Training — Subjects are taught to disengage attention from a certain stimuli
  Arms: Attention Modification Training
Behavioral: No Attention Modification Training — Subjects are exposed to two stimuli, but attention is not manipulated in any way
  Arms: No Attention Modification Training

SUMMARY:
This study aims to examine the effects of smartphone-based Attention-Bias Modification Training (ABMT) in chronic pain participants.

ELIGIBILITY:
Inclusion Criteria:

* existing chronic pain condition

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 1 hour
  questionnaire (numerical pain rating scale)

SECONDARY OUTCOMES:
pain interference | 1 hour
  questionnaire (pain interference scale)

CONTACTS AND LOCATIONS:
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided